CLINICAL TRIAL: NCT04806100
Title: Effects of Malleo-Lok Stiffness on Lower Limb Mechanics
Acronym: MalleoLokStiff
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Jason Wilken, Associate Professor, University of Iowa
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 202004402
Record Dates: First submitted 2021-03-11; First posted 2021-03-19 (Actual); Results first posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-05

CONDITIONS: Adult ALL; Healthy
Keywords: Gait Analysis; Ankle Foot Orthosis; Carbon Fiber; Biomechanics
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Intervention Model Description: All participants will be tested wearing no brace and two braces of differing stiffness's. The testing order will be randomized for each participant to prevent testing order from influencing study results.
Who Masked: Participant
Masking Description: Participants will be blinded to the stiffness of each brace. Braces will be labeled A and B, with stiffness only known by research staff.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (6):
- Compliant, NoCDO, Stiff (Experimental): Participants will be tested while wearing a moderate stiffness device (Compliant), then while wearing no brace (NoCDO), then while wearing a stiff device (Stiff).
  Interventions: Device: Malleo-Lok
- Compliant, Stiff, NoCDO (Experimental): Participants will be tested while wearing a moderate stiffness device (Compliant), then while wearing a stiff device (Stiff), then while wearing no brace (NoCDO).
  Interventions: Device: Malleo-Lok
- NoCDO, Compliant, Stiff (Experimental): Participants will be tested while wearing no brace (NoCDO), then a moderate stiffness device (Compliant), then while wearing a stiff device (Stiff).
  Interventions: Device: Malleo-Lok
- NoCDO, Stiff, Compliant (Experimental): Participants will be tested while wearing no brace (NoCDO), then while wearing a stiff device (Stiff), then while wearing a moderate stiffness device (Compliant).
  Interventions: Device: Malleo-Lok
- Stiff, Compliant, NoCDO (Experimental): Participants will be tested while wearing a stiff device (Stiff), then while wearing a moderate stiffness device (Compliant), then while wearing no brace (NoCDO).
  Interventions: Device: Malleo-Lok
- Stiff, NoCDO, Compliant (Experimental): Participants will be tested while wearing a stiff device (Stiff), then while wearing no brace (NoCDO), then while wearing a moderate stiffness device (Compliant).
  Interventions: Device: Malleo-Lok

INTERVENTIONS:
Device: Malleo-Lok — The Malleo-Lok is a novel, low-profile carbon fiber device with two laterally positioned struts aligned in the sagittal plane.
  Other Names: Ankle Foot Orthosis; Carbon Fiber Custom Dynamic Orthosis

SUMMARY:
The primary purpose of this research study is to determine if the stiffness of a commercially available ankle foot orthosis (Malleo-Lok, Bio-Mechanical Composites, Des Moines IA) impacts gait biomechanics and overall joint level stiffness. Previously published research suggests that AFO stiffness can affect gait biomechanics and patient preference. However, previous studies have focused on traditional posterior strut devices with the strut aligned in the frontal plane to allow sagittal plane deflection. The Malleo-Lok is a novel, low-profile carbon fiber device with two laterally positioned struts aligned in the sagittal plane. The proposed study will provide insight that can be used by certified prosthetists orthotists (CPOs), physical therapists, and physicians to select the device that bests meets their patients' needs.

DETAILED DESCRIPTION:
Healthy adult individuals will be invited to participate in this study, at the University of Iowa, that involves one visit lasting 3-4 hours. The primary purpose of this work is to determine the effects of Malleo-Lok stiffness on gait biomechanics and ankle joint stiffness. Previous work has highlighted the effects of ankle foot orthosis stiffness on gait using devices with a traditional single posterior strut opposed to the Malleo-Lok, which has two laterally positioned struts. Orthosis stiffness is an important factor to consider during device prescription and manufacturing. The ability to tune overall joint level stiffness by determining the combined effects of biological limb stiffness and orthosis stiffness will enhance precision medicine when treating individuals who require an orthosis for daily activities. The secondary purpose of this research study is to determine the within session repeatability of a novel approach for in-vivo AFO stiffness testing. AFO stiffness testing is typically performed using mechanical testing systems without accounting for the interaction of the individual and the device.

During the visit to the University of Iowa campus participants will review a list of inclusion and exclusion criteria to determine their eligibility for this study. Eligible participants will review an informed consent document and have the chance to ask any questions they may have. Study staff will thoroughly explain the informed consent document and answer all questions. Upon signing the informed consent document study activities will begin. Participants will complete all study activities wearing no brace and two braces of differing stiffness's. Anthropometric and demographic information will be collected from each participant. The investigators will also use a motion capture system to evaluate gait biomechanics and ankle joint stiffness. Participants will walk at a self-selected and a controlled speed to evaluate gait biomechanics, and will stand in the motion capture system and bring their knee forward over the foot to evaluate ankle joint stiffness. Participants will be provided visual feedback of muscle activity to minimize lower limb muscle activity during ankle stiffness testing.

Results from the proposed study will provide information about the effects of orthosis stiffness on gait biomechanics and ankle joint stiffness. Study results will be made available to clinicians to use when prescribing and fitting individuals with ankle foot orthoses.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 45
* Healthy without current complaint of lower extremity pain, spine pain, open wounds or active infections, or medical or neuromusculoskeletal disorders that have limited their participation in work or exercise in the last 6 months
* Able to hop without pain
* Able to perform a full squat without pain
* Ability to speak and understand English

Exclusion Criteria:

* Diagnosed with a moderate or severe brain injury
* Lower extremity injury resulting in surgery or limiting function for greater than 6 weeks
* Injuries that would limit performance in this study
* History of recurrent ankle sprains or chronic ankle instability
* Diagnosed with a physical or psychological condition that would preclude functional testing (e.g. cardiac condition, clotting disorder, pulmonary condition)
* Uncorrected visual or hearing impairment(s)
* Require use of an assistive device
* Unhealed wounds (cuts/abrasions) that would prevent AFO use
* BMI > 35
* Pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason M Wilken, PT, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants completed study activities in each of the experimental conditions (NoCDO, Compliant, Stiff) in a randomized order.
Period: Overall Study
Arm/Group | Compliant, NoCDO, Stiff | Compliant, Stiff, NoCDO | NoCDO, Compliant, Stiff | NoCDO, Stiff, Compliant | Stiff, Compliant, NoCDO | Stiff, NoCDO, Compliant
Started | 5 | 5 | 3 | 2 | 4 | 1
Completed | 5 | 5 | 3 | 2 | 4 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants completed study activities in each of the experimental conditions (NoCDO, Compliant, Stiff) in a randomized order.
Groups:
- Total: Total of all reporting groups
Arm/Group | Compliant, NoCDO, Stiff | Compliant, Stiff, NoCDO | NoCDO, Compliant, Stiff | NoCDO, Stiff, Compliant | Stiff, Compliant, NoCDO | Stiff, NoCDO, Compliant | Total
Number analyzed (Participants) | 5 | 5 | 3 | 2 | 4 | 1 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 3 | 2 | 4 | 1 | 20
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.0 (10.6) | 26.0 (5.1) | 28.0 (6.9) | 26.0 (2.8) | 22.5 (2.5) | 27.0 (0.0) | 26.9 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 0 | 4 | 0 | 11
  Male | 3 | 2 | 1 | 2 | 0 | 1 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 1 | 0 | 2
  Not Hispanic or Latino | 5 | 4 | 3 | 2 | 3 | 1 | 18
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 2 | 3 | 1 | 3 | 1 | 13
  More than one race | 0 | 1 | 0 | 1 | 0 | 0 | 2
  Unknown or Not Reported | 2 | 2 | 0 | 0 | 0 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Ankle Joint Stiffness
Description: Ground reaction force and ankle motion data were collected simultaneously using the force measurement and motion capture systems as participants wore no brace (NoCDO), a moderate stiffness orthosis (Compliant) and a stiff orthosis (Stiff) in a randomized order. The ankle motion data was plotted against the ankle moment data and the slope of the corresponding line was the resulting ankle joint stiffness (Nm/degree).
Time Frame: In-vivo ankle joint stiffness was measured for each condition before and after short bouts of walking (~15-20 minutes).
Population: All participants completed all study activities (in-vivo ankle stiffness testing, walking, questionnaires) for each of the experimental conditions (NoCDO, Compliant, Stiff) in a randomized order.
Measure: Mean (Standard Deviation); unit: Nm/degree
Groups:
- NoCDO: Participants will be tested while wearing no brace (NoCDO)
- Compliant: Participants will be tested while wearing a moderate stiffness orthosis (Compliant)
- Stiff: Participants will be tested while wearing a stiff orthosis (Stiff).
Arm/Group | NoCDO | Compliant | Stiff
Number analyzed (Participants) | 20 | 20 | 20
Nm/degree | 0.62 (0.32) | 0.97 (0.34) | 0.98 (0.34)

2. Primary Outcome: Ankle Joint Power
Description: Peak ankle joint push-off power (W/kg) was calculated during gait and normalized to participant body weight as participants wore no brace (NoCDO), a moderate stiffness orthosis (Compliant) and a stiff orthosis (Stiff) in a randomized order.
Time Frame: Ankle joint power was measured for each condition during short bouts of walking (~15-20 minutes).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: W/kg
Arm/Group | NoCDO | Compliant | Stiff
Number analyzed (Participants) | 20 | 20 | 20
W/kg | 2.8 (0.5) | 2.2 (0.4) | 2.1 (0.3)

3. Primary Outcome: Ankle Joint Moment
Description: Peak ankle plantarflexion moment (Nm/kg) was calculated during gait and normalized to participant body weight as participants wore no brace (NoCDO), a moderate stiffness orthosis (Compliant) and a stiff orthosis (Stiff) in a randomized order.
Time Frame: Ankle joint moment was measured for each condition during short bouts of walking (~15-20 minutes).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Nm/kg
Arm/Group | NoCDO | Compliant | Stiff
Number analyzed (Participants) | 20 | 20 | 20
Nm/kg | 1.4 (0.1) | 1.3 (0.1) | 1.3 (0.1)

4. Secondary Outcome: Numerical Pain Rating Scale
Description: Participants were asked to rate their pain on a standard 11-point numerical pain rating scale, in which 0 = no pain and 10 = worst pain imaginable. Participants were asked to rate their pain after completing testing in no brace (NoCDO), a moderate stiffness orthosis (Compliant) and a stiff orthosis (Stiff) in a randomized order.
Time Frame: Participants were asked to rate their pain after completing in-vivo ankle stiffness testing and walking trials in all conditions.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NoCDO | Compliant | Stiff
Number analyzed (Participants) | 20 | 20 | 20
score on a scale | 0.1 (0.2) | 0.2 (0.5) | 0.2 (0.5)

5. Secondary Outcome: Modified Socket Comfort Score: Comfort
Description: Study participants were asked to rank the smoothness of each orthosis on a scale from 0-10 where 0 = least smooth and 10 = most smooth orthosis. Participants were asked to rate the comfort of each orthosis after completing testing in a moderate stiffness orthosis (Compliant) and a stiff orthosis (Stiff) in a randomized order.
Time Frame: Participants were asked to rate their comfort after completing in-vivo ankle stiffness testing and walking trials in Compliant and Stiff conditions.
Population: All participants completed all study activities (in-vivo ankle stiffness testing, walking, questionnaires) for each of the experimental conditions (NoCDO, Compliant, Stiff) in a randomized order. The modified socket comfort score does not apply to walking without an orthosis, so was not assessed for the NoCDO condition.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Compliant | Stiff
Number analyzed (Participants) | 20 | 20
score on a scale | 7.5 (1.7) | 8.0 (1.6)

6. Secondary Outcome: Modified Socket Comfort Score: Smoothness
Description: Study participants were asked to rank the smoothness of each orthosis on a scale from 0-10 where 0 = least smooth and 10 = most smooth orthosis. Participants were asked to rate the smoothness of each orthosis after completing testing in a moderate stiffness orthosis (Compliant) and a stiff orthosis (Stiff) in a randomized order.
Time Frame: Participants were asked to rate the orthosis smoothness after completing in-vivo ankle stiffness testing and walking trials in Compliant and Stiff conditions.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Compliant | Stiff
Number analyzed (Participants) | 20 | 20
score on a scale | 7.8 (1.7) | 7.7 (2.0)

7. Other Pre Specified Outcome: Center of Pressure Velocity Magnitude
Description: Magnitude of peak center of pressure velocity (m/s) during gait.
Time Frame: Baseline
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Center of Pressure Velocity Timing
Description: Timing of peak center of pressure velocity (percent stance) during gait.
Time Frame: Baseline
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Soleus Muscle Activity (Electromyography)
Description: Electromyography of soleus activity during in-vivo ankle stiffness testing was used as visual feedback for participants during testing.
Time Frame: Baseline
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Medial Gastrocnemius Muscle Activity (Electromyography)
Description: Electromyography of medial gastrocnemius activity during in-vivo ankle stiffness testing was used as visual feedback for participants during testing.
Time Frame: Baseline
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Tibialis Anterior Muscle Activity (Electromyography)
Description: Electromyography of tibialis anterior activity during in-vivo ankle stiffness testing was used as visual feedback for participants during testing.
Time Frame: Baseline
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Peroneus Longus Muscle Activity (Electromyography)
Description: Electromyography of peroneus longus activity during in-vivo ankle stiffness testing was used as visual feedback for participants during testing.
Time Frame: Baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Study participants were asked to indicate any adverse events throughout the duration of the study visit. After completion of the study visit participants were also asked to call or email the research team if any adverse events related to the study occurred after the study visit (up to ~12 months after the visit).
Arm/Group | NoCDO | Compliant | Stiff
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-11): https://cdn.clinicaltrials.gov/large-docs/00/NCT04806100/Prot_SAP_001.pdf